CLINICAL TRIAL: NCT05555108
Title: Mindfulness and Compassive Acceptance for Chronic Insomnia in Comparison With CBT
Acronym: ACTCOM-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Mariana Miller-Mendes, PhD fellowship at Center for Research in Neuropsychology and Cognitive Bebavioral Intervention (CINEICC), University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFRH/BD/147556/2019
Record Dates: First submitted 2022-05-30; First posted 2022-09-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Insomnia; CBT
Keywords: Chronic Insomnia; CBT-I; ACT; Compassion
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTCOM-I Intervention (Experimental)
  Interventions: Behavioral: ACTCOM-I Intervention
- Standard CBT-I Intervention (Active Comparator)
  Interventions: Behavioral: Standard CBT-I Intervention

INTERVENTIONS:
Behavioral: ACTCOM-I Intervention — ACTCOM-I s an individual treatment protocol based on Acceptance and Commitment Therapy (ACT) with targeted behavioral components for insomnia treatment and a specific focus on selfcompassion as a protector for sleep disturbance.
  Arms: ACTCOM-I Intervention
Behavioral: Standard CBT-I Intervention — Standard CBT-I treatment for chronic insomnia. Treatment protocol adapted from Morin's protocol (1993)
  Arms: Standard CBT-I Intervention

SUMMARY:
The main aim of this study is to test the efficacy of a Compassive Acceptance Intervention protocol (developed by the research team) for Chronic Insomnia in comparison with the standard treatment (CBT-I).

ELIGIBILITY:
Inclusion Criteria:

* Insomnia Diagnosis (ICSD-3; DSM-5)

Exclusion Criteria:

* Comorbidity with severe psychiatric/psychological disorder (e.g. severe depression; psychotic disorder)
* Comorbidity with other untreated sleep disorder
* Altered Sleep patterns due to factors different from insomnia (e.g. shift-work; pregnancy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Change in insomnia severity scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Insomnia severity assessed by the Insomnia Severity Index (ISI). The ISI is a 7-item self-report questionnaire that evaluates the nature, severity, and impact of insomnia. Scores range from 0 to 28 points with higher scores indicating more severe insomnia symptoms.

SECONDARY OUTCOMES:
Change in pre-sleep arousal scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Pre-sleep arousal assessed by the Pre-Sleep Arousal Scale (PSAS). The PSAS is a 16-item self-report questionnaire that evaluates symptoms of arousal at bedtime. Eight items evaluate symptoms of cognitive arousal and eight evaluate symptoms of somatic arousal experienced when attempting to fall asleep. Scores range from 8 to 40 in each subscale, where higher scores indicate greater activation.
Change in sleep effort scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Sleep effort assessed by the Glasgow Sleep Effort Scale (GSES). The GSES is a 7-item self-report questionnaire that evaluates the presence of a state of sleep effort. Scores range from 0 to 14 where higher scores indicate greater effort to sleep
Change in dysfunctional beliefs and attitudes about sleep scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Dysfunctional beliefs and attitudes about sleep assessed by the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS). The DBAS is a 30-item self-report questionnaire that addresses several beliefs and attitudes about sleep and insomnia. A global score is found by averaging scores on all items, with higher scores indicating more dysfunctional beliefs and attitudes about sleep.
Change in anxiety and depression symptoms scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Anxiety and depression symptoms assessed by the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item self-report questionnaire of which 7 items assess depression and 7 items assess anxiety. Scores range from 0 to 21 for each subscale where higher scores denote higher distress (anxiety and depression).
Change in positive and negative affect scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Assessment of affect using the PANAS Portuguese Short Version (PANAS-VRP). The PANAS-VRP is a 10-item self-report questionnaire of which 5 items evaluate positive affect and 5 items evaluate negative affect. Scores range from 5 to 25 for each subscale where higher scores indicate high positive and negative affect, for each subscale respectively.
Change in trait mindfulness scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Assessment of trait mindfulness using the Five Facet Mindfulness Questionnaire (FFMQ). The FFMQ is a 39-item self-report questionnaire evaluating the trait-like tendency to be mindful in daily life. The scale provides a global mindfulness score (sum of each facet score) and comprises five related facets (observing; describing; acting with awareness; nonjudging; nonreactivity). Facet scores range from 8-40, except for the nonreactivity facet, which ranges from 7-35. Higher scores indicate higher mindfulness trait.
Change in psychological flexibility scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Assessment of psychological inflexibility or experiential avoidance using the Acceptance and Action Questionnaire-II (AAQ-II). The AAQ-II is a 7-item self-report questionnaire with total scores ranging from 7 to 49 where higher scores indicate higher levels of psychological inflexibility.
Change in cognitive fusion scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Assessment of the process of cognitive fusion using the Cognitive Fusion Questionnaire (CFQ). The CFQ is a 7-item self-report questionnaire that evaluates the degree to which people tend to fuse with their thoughts. Scores range from 7 to 49 points, where higher scores indicate higher levels of cognitive fusion.
Change in personal values enactment scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Assessment of one's engagement in valued action (personal values enactment) using the Valuing Questionnaire (VQ). The VQ is a 10-item self-report questionnaire that evaluates how consistently an individual is living according with their chosen values. The scale measures two constructs - progress and obstruction - and each subscale is scored from 0 to 30 points. On the progress subscale, higher scores indicate higher valued based action and, on the obstruction subscale, higher scores denote higher interference with acting according to one's values.
Change in self-compassion scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Assessment of self-compassion using the Self-Compassion Scale (SCS). The SCS is a 26-item self-report questionnaire that evaluates the capacity for self-compassion through six subscales (Self-Kindness; Self-Judgment; Common Humanity; Isolation; Mindfulness; Over-identification). Total scores range from 26 to 130 points. Higher scores indicate higher self-compassion for total scores and subscale scores.
Change in Quality of life scores | Baseline (2 weeks prior the start of treatment), post-treatment (2 weeks after the 10th session - treatment completion), 3 months after treatment completion, 6 months after treatment completion
  Assessment of individual facets relating to quality of life using the World Health Organization Quality Of Life Scale (WHOQOL-BREF). The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items). Total scores range from 26 to 130 points. Higher scores indicate better satisfaction with quality of life on total score and subscale scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Medicina do Sono do Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal